CLINICAL TRIAL: NCT07139951
Title: Prophylactic Hyperthermic IntraperitOneal Chemotherapy (p-HIPEC) for pRevention of perItONeal Recurrence in Gastric Cancer: MC240402 (HORIZON) Trial
Brief Title: Hyperthermic Intraperitoneal Chemotherapy With Cisplatin and Paclitaxel for the Treatment of Patients With Gastric and Gastroesophageal Junction Adenocarcinoma at High Risk of Peritoneal Recurrence
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC240402; NCI-2025-05845 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-013133 (Other: Mayo Clinic Institutional Review Board); MC240402 (Other: Mayo Clinic)
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage I Gastric Cancer AJCC v8; Clinical Stage I Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage II Gastric Cancer AJCC v8; Clinical Stage II Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Biopsy; Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Hyperthermic Intraperitoneal Chemotherapy; Laparoscopy; Lymph Node Excision; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (p-HIPEC, cisplatin, paclitaxel) (Experimental): Patients undergo gastrectomy with reconstruction per surgeon discretion and D2 lymphadenectomy and receive p-HIPEC with cisplatin and paclitaxel intraperitoneal (IP) over 90 minutes on study. Patients also undergo blood sample collection and PET/CT or PET/MRI throughout the study, as well as laparoscopy with biopsy during screening.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Hyperthermic Intraperitoneal Chemotherapy; Procedure: Laparoscopy; Procedure: Lymphadenectomy; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo laparoscopy with biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IP
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Hyperthermic Intraperitoneal Chemotherapy — Given p-HIPEC
  Other Names: HIPEC
Procedure: Laparoscopy — Undergo laparoscopy with biopsy
  Other Names: LP
Procedure: Lymphadenectomy — Undergo D2 lymphadenectomy
  Other Names: excision of the lymph node; Lymph Node Dissection; Lymph Node Excision
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IP
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Positron Emission Tomography — Undergo PET/CT or PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Surgical Procedure — Undergo gastrectomy and reconstruction
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase II trial tests how well concentrating heated (hyperthermic) chemotherapy in the area that contains the abdominal organs (intraperitoneal [IP]) at the time of surgery works in treating patients with gastric or gastroesophageal junction adenocarcinoma at high risk of the cancer coming back to the abdominal cavity (peritoneal) after a period of improvement (recurrence). Recurrence in the peritoneum often occurs within the first 18 months after surgery. This is thought to be due to tumor cells that may scatter and spread during surgery. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Paclitaxel is in a class of medications called antimicrotubule agents. It stops tumor cells from growing and dividing and may kill them. Paclitaxel alone and in combination with other chemotherapy agents have been shown to be effective treatments for gastric tumors. However, systemic delivery of these drugs has not been shown to be effective in treating peritoneal metastasis. Hyperthermic intraperitoneal chemotherapy (HIPEC) is a procedure that involves the infusion of a heated chemotherapy solution, such as cisplatin and paclitaxel, that circulates into the abdominal cavity. Giving HIPEC with cisplatin and paclitaxel at the time of surgery may reduce peritoneal recurrence in patients with gastric or gastroesophageal junction adenocarcinoma at high risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years
* Histological confirmation of adenocarcinoma of the stomach or gastroesophageal junction (GEJ) (Siewert type II or III)
* Tumor index (TI) ≥ 90 (T stage multiplied by the largest tumor diameter in mm on endoscopic ultrasound [EUS]). Patients with linitus plastica automatically have TI ≥ 90
* Hemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1000/mm^3
* Platelet count ≥ 75,000/mm^3
* Calculated creatinine clearance ≥ 60 ml/min using the Cockcroft-Gault formula
* No radiographic or histological evidence of distant metastasis
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an agent that has known genotoxic, mutagenic, and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential and persons able to father a child who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Renal insufficiency (estimated glomerular filtration rate [eGFR] < 60)
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Active second malignancy currently receiving systemic treatment ≤ 6 months prior to pre-registration
* History of myocardial infarction ≤ 6 months prior to pre-registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2031-11-03 (Estimated)

PRIMARY OUTCOMES:
Peritoneal Recurrence-free Survival | Up to 18 months
  Patients will be followed in active surveillance with biomarkers (CEA and CA 19-9) and cross-sectional imaging of the chest, abdomen and pelvis. Only non-lymphatic, non-peranastomotic, and non-visceral intra-abdominal metastasis will be considered peritoneal metastasis. Ovarian metastasis will be considered peritoneal metastasis for this trial.

SECONDARY OUTCOMES:
Safety and Tolerability (Adverse Events) | Up to 45 days after study treatment
  Safety and tolerability will be determined by incidence of adverse events (AEs), specifically the incidence of grade 3 neutropenia and thrombocytopenia. AEs will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The incidence of acute kidney injury will be defined by the glomerular filtration rate (GFR) criteria of the Risk, Injury, Failure, Loss of kidney function and End-stage kidney disease (RIFLE) classification.
Recurrence-free Survival | Up to 5 years
  Recurrence-free survival (RFS) is defined as the time from study entry to the first of either disease progression or death due to any cause. Any radiographic, endoscopic or biopsy proven recurrence of cancer will count as disease recurrence.
Overall Survival | 3 years and 5 years
  Overall survival (OS) is defined as the time from date of study entry to date of death or last follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Travis E. Grotz, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials